CLINICAL TRIAL: NCT02894242
Title: The Evaluation of a Nasal Pillows Mask for the Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-197
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F&P Deimos Nasal Pillows Mask (Experimental): Participants to use nasal pillows mask in-home for 2 weeks.
  Interventions: Device: F&P Deimos Nasal Pillows Mask

INTERVENTIONS:
Device: F&P Deimos Nasal Pillows Mask — Investigative Nasal Pillows Mask to be used for OSA therapy
  Other Names: Deimos Mask

SUMMARY:
This investigation is designed to evaluate the performance as well as the patients overall acceptance of the mask.

DETAILED DESCRIPTION:
A minimum of 20 OSA participants who currently use a nasal pillows mask will be recruited for the trial. Participant will be on the trial for three weeks - first week will be a collection of Positive Airway Pressure (PAP) baseline data on the participant's usual mask. The participant will then use the trial mask in-home for 2 weeks. There is also an option of a two month extension if the participant wish to continue on the trial mask.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* Apnea hypopnea Index (AHI)≥ 5 on diagnostic night
* Prescribed PAP for OSA
* Existing nasal pillows user

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness
* Anatomical or physiological conditions making automatic positive airway pressure (APAP) therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency
* Current diagnosis of carbon dioxide (CO2) retention
* Pregnant or may think they are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Ease of use | 2 weeks in home
  Subjective questionnaire
Acceptability | 2 weeks in home
  Subjective questionnaire

SECONDARY OUTCOMES:
Objective leak data | 2 weeks in home
  Obtained from participants' device

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Gunson, Bsc PgDip, Principal Investigator — Sponsor Employee
Locations (2):
- New Zealand (2):
  - Fisher and Paykel Healthcare, Auckland
  - Hawkes Bay Fallen Soldiers' Memorial Hospital, Hastings

IPD SHARING:
Plan to Share IPD: No
For product development purposes only. Data will be deidentified.